CLINICAL TRIAL: NCT00716573
Title: COREV : A Multi-center, Randomized, Open-label Study Evaluating the Efficacy on Renal Function of Everolimus in Heart Transplant Recipients With Established Chronic Renal Failure
Brief Title: Efficacy Study of Everolimus on Renal Function in Heart Transplant Recipients With Established Chronic Renal Failure
Acronym: COREV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007.495
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Cardiac Transplantation; Chronic Renal Insufficiency
Keywords: Cardiac transplantation; Chronic renal insufficiency; Everolimus
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Introduction of everolimus associated with CNI (ciclosporin or tacrolimus) reduction (50%) to the current immunosuppression schedule
  Interventions: Drug: everolimus
- 2 (No Intervention): Maintain of their current immunosuppressive therapy

INTERVENTIONS:
Drug: everolimus — 0,75 mg bid, 24 months
  Other Names: Certican
  Arms: 1

SUMMARY:
After transplantation, renal impairment, incidence and progression of atherosclerosis lead to modification of immunosuppressive regimens, as switch, reduction or discontinuation of CNI and/or introduction of everolimus. The risk or benefits of these strategies were not clearly evaluated by specific clinical trials.

This study is specifically designed for evaluating the impact of everolimus introduction, with calcineurin dose reduction, at less one year after cardiac transplantation, on renal and clinical outcomes, specially on :

* Renal function improvement
* Vasculopathy and major cardiac event reduction
* Maintenance of immunosuppressive efficacy

ELIGIBILITY:
Inclusion Criteria:

* Male or female cardiac recipients over 18 years old
* First or second heart transplant, more than one year following surgery
* Patients with renal failure assessed by cGFR 30 to 60 ml/min/1,73m² calculated by MDRD4 formula
* Patients volunteer to participate in the study, with a written informed consent signed
* Affiliation to a national health insurance program

Exclusion Criteria:

* Current CNI-free immunosuppressive regimen
* Patients currently or previously treated with a mTOR inhibitor any time prior randomization
* Patients who are recipients for a multiple solid organ transplant
* Treated acute rejection episode within three months prior randomization
* Congestive heart failure (NYHA class III or IV) and/or VEF < 30 % and/or patient waiting for a re-transplantation
* Scheduled surgical intervention
* Platelet count < 50 G/l
* Severe hepatic insufficiency (SGPT and/or SGOT > 3N)
* Major lipidic profile abnormalities (total cholesterol > 3g/l and/or TG > 5g/l)
* Proteinuria/creatinuria > 0,08 g/mmol
* Severe renal failure attested by cGFR < 30 ml/min/1.73m² (MDRD4)
* History of Hypersensitivity to everolimus, sirolimus or excipients
* History of Hypersensitivity to macrolides
* Pregnancy and breast feeding
* Childbearing age women without efficient contraception
* Law protected patients
* Patients in emergency unable to express their consent
* History of Hypersensitivity to cyclosporine or St-John's wort, stiripentol, bosentan, rosuvastatin
* History of Hypersensitivity to tacrolimus, macrolides or excipients
* History of Hypersensitivity to azathioprine
* History of Hypersensitivity to mycophénolate mofetil or excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-09-16 (Actual); Primary Completion 2014-04-17 (Actual); Study Completion 2014-04-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of the renal function, at 12 months after everolimus introduction and doses of anticalcineurins decrease. | 12 months

SECONDARY OUTCOMES:
Evaluation of the benefit of everolimus introduction on renal function at 24 months | 24 months
Evaluation of the benefit of everolimus introduction on incidence of Major Adverse Cardiac Events (MACEs) | 24 months
Evaluation of the benefit of everolimus introduction on incidence of cardiovascular risk factor (Arterial Tension, diabetes, dyslipidemia, proteinuria) | 24 months
Evaluation of the benefit of everolimus introduction on incidence of treatment withdrawals | 24 months
Evaluation of the benefit of everolimus introduction on incidence of treated acute rejection | 24 months
Evaluation of the benefit of everolimus introduction on safety | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pascale BOISSONNAT, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France